CLINICAL TRIAL: NCT01603472
Title: Markers of Parenteral Nutrition (PN) Associated Metabolic Bone Disease in Children on Long-Term PN for Intestinal Failure.
Brief Title: Markers of Bone Disease in Children on Parenteral Nutrition
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Rare Disease Foundation, Vancouver, Canada (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Academic &Clinical Specialist, Project Investigator, The Hospital for Sick Children
Other Study IDs: 1000028242
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Metabolic Bone Disease
Keywords: pediatric; parenteral nutrition; bone disease; long-term PN
MeSH Terms: conditions — Bone Diseases, Metabolic; Hyperphagia; Bone Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects on Parenteral Nutrition: cases are those on Parenteral Nutrition >6 weeks for intestinal failure.
- Subjects not on Parenteral Nutrion: Controls are those who have never been on PN but can be fed via a feeding tube

SUMMARY:
Parenteral nutrition (PN) is the provision of nutrients via the intravenous route. Parenteral nutrition associated metabolic bone disease (MBD) was first described in children in the 1980s. Since then, there has been little to no research into the underlying relationship and as a result, little evidence on which to base clinical care. In adults, MBD is associated with increased fractures. At the Hospital for Sick children in Toronto, an intestinal failure program has been set up since 2003. This is the only intestinal failure program in Canada and receives country wide referrals. Most of the patients have short bowel syndrome (SBS) and require PN for prolonged periods, or for life. About 90% of these patients have MBD, and some have had bone fractures. An understanding of the etiology of MBD would provide information to guide care, and prevent this condition. Funding for this area of research however is challenging because intestinal failure requiring long term PN is a rare condition, accounting for approximately 200 - 300 children in all of Canada. The goal of this study therefore is to gather pilot data on markers of MBD in children on long term PN, and to compare these markers to age and gender matched control patients who are fed by mouth or feeding tube. The information gathered from this study will help us begin to understand what is actually happening in the bones of children on long term PN and will form the basis for future studies and improved clinical care.

ELIGIBILITY:
INCLUSION CRITERIA:

For Cases on Long-term PN:

1. On PN for ≥ 6 consecutive weeks
2. Willingness to participate in the study

For Control Subjects:

1. Healthy as assessed by history and physical exam.
2. Growing normally
3. Are not on medications known to affect bone metabolism eg. Corticosteroids.
4. Never received PN in the past

EXCLUSION CRITERIA:

For Cases on Long-term PN

1. Patients who are on PN for shorter than 6 weeks
2. Patients on hemodialysis

For Control Subjects

1. Subjects who are not able to be matched to a case/subject on long-term PN for age and gender
2. Positive history of fractures
3. Subjects who are unable to participate because of fear of giving blood or unable to come to the hospital for sick children for blood draws.

Ages: 6 Weeks to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children on long term PN and childen not on PN.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
serum osteocalcin | Over 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada